CLINICAL TRIAL: NCT01535560
Title: Safety and Efficacy Evaluation of Topical AL-60371 Otic Suspension, 0.3% in the Treatment of Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-019
Record Dates: First submitted 2012-02-15; First posted 2012-02-17 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-10

CONDITIONS: Acute Otitis Externa
Keywords: Acute otitis externa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-60371 (Experimental): AL-60371, 0.3% otic suspension, 4 drops in the affected ear(s) twice daily for 7 days
  Interventions: Drug: AL-60371, 0.3% otic suspension
- Vehicle (Placebo Comparator): AL-60371 Vehicle, 4 drops in the affected ear(s) twice daily for 7 days
  Interventions: Drug: AL-60371 Vehicle

INTERVENTIONS:
Drug: AL-60371, 0.3% otic suspension — Investigational otic suspension intended for the treatment of acute otitis externa
  Arms: AL-60371
Drug: AL-60371 Vehicle — Inactive ingredients used as placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study was to demonstrate superiority of AL-60371 relative to Vehicle based on clinical cures at test-of-cure (TOC) for the treatment of acute otitis externa (AOE).

DETAILED DESCRIPTION:
Participants or legal guardians completed a telephone diary twice daily to record assessments of ear pain, ear medication use, and impact of ear pain on sleep and other daily activities.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of age.
* Clinical diagnosis of acute otitis externa (AOE) based on clinical observation and of presumed bacterial origin in at least one ear.
* Combined numerical score of ≥4 in at least one affected ear at the Day 1 exam for tenderness, erythema, and edema.
* Agree to refrain from water immersion of the ears during the conduct of the entire study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Duration of signs or symptoms of AOE greater than 28 days in the affected ear(s) as reported by patient or parent/guardian.
* Presence of a tympanostomy tube or perforated tympanic membrane in the affected ear(s).
* Clinically diagnosed otic disease other than AOE (eg, malignant otitis externa) in the affected ear(s).
* Known or suspected ear infection of yeast, fungal or mycobacterial origin in the affected ear(s).
* Prior otologic surgery within 6 months of study entry in the affected ear(s).
* Known or suspected allergy or hypersensitivity to quinolones or other ingredients present in the medications to be used in the study.
* Patients who use ear plugs, head phones or ear buds and are unwilling to discontinue their use during the study period.
* Other protocol-defined exclusion criteria may apply.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Schieb, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 53 investigational centers located in the United States, Puerto Rico, and Canada.
Pre-assignment Details: Of the 589 participants enrolled, 40 were exited from the study as screen failures prior to randomization. This reporting group includes all randomized participants.
Period: Overall Study
Arm/Group | AL-60371 | Vehicle
Started | 274 | 275
Completed | 237 | 179
Not Completed | 37 | 96
Not completed — Adverse Event | 12 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Subj Decision Unrel to an Adverse Event | 3 | 1
Not completed — Treatment Failure | 21 | 83
Not completed — Other | 0 | 1
Not completed — Randomized in Error | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized participants who received the study drug (ie, 548). Note: 1 participant in the Vehicle arm was randomized in error and did not receive the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-60371 | Vehicle | Total
Number analyzed (Participants) | 274 | 274 | 548
Age, Customized [Number; unit: Participants]
  Infants and Toddlers (28 days to 23 months) | 0 | 1 | 1
  Children (2 to 11 years) | 130 | 120 | 250
  Adolescents (12 to 17 years) | 56 | 62 | 118
  Adults (18 to 64 years) | 80 | 87 | 167
  Elderly (≥ 65 years) | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 170 | 318
  Male | 126 | 104 | 230

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Clinical Cures at the Day 11 (TOC) Visit
Description: An otoscopic exam was conducted by the physician. Clinical cure was considered attained if the sum of the numerical scores of the 3 signs and symptoms of AOE (tenderness, erythema, and edema) was 0 at Day 11. Proportion of patients is reported as percentage of participants.
Time Frame: Day 11
Population: This reporting group includes the pathogen positive patients of the intent-to-treat (ITT) analysis set, ie. all patients who received study drug and were pathogen positive in the study ear at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | AL-60371 | Vehicle
Number analyzed (Participants) | 147 | 130
Percentage of participants | 68.7 | 40.0

2. Secondary Outcome: Proportion of Patients With Microbiological Successes at the Day 11 (TOC) Visit
Description: Microbiological success was considered attained if all pre-therapy bacteria were absent from the exit otic specimen. The presence of fungi and/or yeast was not considered in the determination of microbiological success. Proportion of patients is reported as a percentage of participants.
Time Frame: Day 11
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AL-60371 | Vehicle
Number analyzed (Participants) | 147 | 130
Percentage of participants | 66.0 | 11.5

3. Secondary Outcome: Median Time (in Days) to Cessation of Ear Pain as Reported by the Patient or Parent/Legal Guadian Via the Telephone Diary
Description: Cessation of ear pain was defined as occurring the first time point that ear pain was absent (morning or evening) and did not reoccur in any subsequent diary entries.
Time Frame: Time to event (Day 1 to Day 11)
Population: This reporting group includes the pathogen positive patients of the intent-to-treat (ITT) analysis set, ie. all patients who received study drug and were pathogen positive in the study ear at baseline, minus missing responses.
Measure: Median (Standard Error); unit: Days
Arm/Group | AL-60371 | Vehicle
Number analyzed (Participants) | 138 | 125
Days | 3.0 (0.2) | 6.5 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (6 months).
Description: This reporting group includes all participants who received study drug. Adverse events were obtained as solicited comments from the study patients and as observations by the study investigator.
Arm/Group | AL-60371 | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/274 | 0/274
Other Adverse Events (participants affected / at risk) | 0/274 | 0/274

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.